CLINICAL TRIAL: NCT03866278
Title: Characterizing the Electroencephalogram Signature of Fentanyl During Induction of General Anesthesia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick L. Purdon, Associate Professor of Anesthesia, Massachusetts General Hospital
Other Study IDs: 2018P000383; 5R21DA048323-02 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2019-03-07 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia
Keywords: Opiate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While historically anesthesiologists rely on pharmacokinetics to track the loss of consciousness, new research in anesthesiology has identified the salient features of the electroencephalogram (EEG) that correlate to states of sedation and unconsciousness induced by different anesthetic drugs. While the EEG features of many sedative-hypnotic anesthetics have been well- characterized, the opioid analgesic drugs have not been analyzed in detail in this way. A characterization of the EEG signatures of opioid analgesic drugs could be useful in monitoring and titrating the effects of these drugs.

DETAILED DESCRIPTION:
Fentanyl is one of the most commonly used opioid analgesic drugs. Prior to induction of general anesthesia, fentanyl is frequently administered to blunt the nociceptive response to intubation. A typical scenario is to administer 2 to 4 mcg/kg of fentanyl first, followed by a sedative hypnotic drug such as propofol to induce general anesthesia. In this study, we propose to administer a total of 4 mcg/kg of fentanyl, administered in 2 boluses, before administering a sedative hypnotic drug. At this dose, fentanyl will serve to blunt nociception during intubation, but will also contribute to intraoperative pain management. During this time, we will record the EEG using standard EEG-based anesthetic monitors that are routinely used in the operating room. We will assess the patient's level of responsiveness using an auditory task and ulnar nerve stimulation. These measurements will allow us to identify the EEG signatures of fentanyl for future use in EEG-based anesthetic monitoring. During this study we will measure EEG and responses to auditory and ulnar nerve stimuli during induction of general anesthesia in surgical patients. The anesthetic will be administered according to a typical sequence in which fentanyl is first administered, followed by a sedative hypnotic drug for induction of general anesthesia. The primary difference is that, in this study, we will record the EEG and response data for a short period of time after initial administration of fentanyl and prior to administration of a sedative hypnotic drug to induce general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

-Undergoing surgery anticipated to take 2 hours or longer

Exclusion Criteria:

* Craniofacial abnormalities
* Allergies to fentanyl, bisulfite, eggs or egg products, latex, soybeans, soybean oil BMI ≤ 30 (kg/m2)
* Known or suspected difficult intubation
* Known or suspected need for rapid sequence induction and intubation
* History of obstructive sleep apnea requiring CPAP
* History of uncontrolled gastroesophageal reflux disease (GERD)
* Opiate use within 24 hours
* History of opiate abuse within 3 years

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Only those patients capable of giving their own consent will be considered for this study. All study subjects will be American Society of Anesthesiologists (ASA) physical status classification P1 to P3. That is, all study subjects will have at most mild to moderate systemic disease.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Only arm of the study. Subjects received an anesthetic dose of fentanyl during induction to general anesthesia while having vitals and frontal electroencephalogram monitored.
Period: Overall Study
Arm/Group | Study Group
Started | 31
Completed | 28
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 31 subjects were enrolled. 25 subjects finished the protocol.
Arm/Group | Study Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — Measure Analysis Population Description: Two subjects were not studied because of scheduling conflicts, and one further was not studied due to withdrawal of consent.
  There were technical problems in three additional subjects that led to data loss: In one subject, we were unable to record the respiratory signals; in another, we were unable to obtain the behavioral responses; and in yet another, the EEG signal was too noisy to analyze.
  years | 54 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two subjects were not studied because of scheduling conflicts, and one further was not studied due to withdrawal of consent.
  There were technical problems in three additional subjects that led to data loss: In one subject, we were unable to record the respiratory signals; in another, we were unable to obtain the behavioral responses; and in yet another, the EEG signal was too noisy to analyze.
  Participants
    Female | 12
    Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two subjects were not studied because of scheduling conflicts, and one further was not studied due to withdrawal of consent.
  There were technical problems in three additional subjects that led to data loss: In one subject, we were unable to record the respiratory signals; in another, we were unable to obtain the behavioral responses; and in yet another, the EEG signal was too noisy to analyze.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 22
    Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two subjects were not studied because of scheduling conflicts, and one further was not studied due to withdrawal of consent.
  There were technical problems in three additional subjects that led to data loss: In one subject, we were unable to record the respiratory signals; in another, we were unable to obtain the behavioral responses; and in yet another, the EEG signal was too noisy to analyze.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 23
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Population: Two subjects were not studied because of scheduling conflicts, and one further was not studied due to withdrawal of consent.
  There were technical problems in three additional subjects that led to data loss: In one subject, we were unable to record the respiratory signals; in another, we were unable to obtain the behavioral responses; and in yet another, the EEG signal was too noisy to analyze.
  participants
    United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Slope of EEG Theta Band Power Over Fentanyl Effect Site Concentration (dB/ng/mL)
Description: We estimated the fentanyl effect site concentration (ESC) in (nanograms/mL) using pharmacokinetic/pharmacodynamic (PK/PD) modeling implemented in StanpumpR. We estimated EEG power using multitaper spectral analysis and calculated the power in decibels (dB) within the theta band (4 - 8 Hz).
  To quantify the relationship between the EEG and fentanyl concentration, we constructed a linear mixed-effects model representing fentanyl concentration as a function of theta power.
Time Frame: Twenty minutes prior to surgery
Measure: Number (95% Confidence Interval); unit: dB / nano gram / mL
Arm/Group | Study Group
Number analyzed (Participants) | 25
dB / nano gram / mL | 0.55 [0.25 to 0.8]

2. Primary Outcome: Slope of Minute Ventilation Index Over Theta Band Power (Index/dB)
Description: Minute ventilation is a physiological term that refers to the total volume of air a person breathes in and out of their lungs in one minute. To calculate this we measured the chest and abdominal expansion and contraction and estimated the instantaneous frequency and instantaneous amplitude. This measure is relative to a baseline minute ventilation defined as "tidal volume" and is therefore a dimensionless number between 0 and 1 where 1 is equivalent to the baseline tidal volume.
  We estimated the EEG power in decibels (dB) within the theta band range (4-8 Hz). To characterize the relationship between "theta band power" and respiratory changes (Minute Ventilation Index) we constructed a mixed-effects model.
Time Frame: Twenty minutes prior to surgery
Measure: Number (95% Confidence Interval); unit: index/dB
Arm/Group | Study Group
Number analyzed (Participants) | 25
index/dB | -1.62 [-2.51 to 0.73]

3. Primary Outcome: Slope of Response Time Over Minute Ventilation Index (Milliseconds/Index)
Description: We measured the response time to auditory stimuli in milliseconds. We measured the changes in Minute Ventilation by estimating the instantaneous frequency and instantaneous amplitude of respiratory inductance bands. This measure is relative to a baseline minute ventilation defined as "tidal volume" and is therefore a dimensionless number between 0 and 1 where 1 is equivalent to the baseline tidal volume.
  We used a linear mixed-effects models to characterize reaction time as a function of minute ventilation index.
Time Frame: Twenty minutes prior to surgery
Measure: Number; unit: milliseconds/index
Arm/Group | Study Group
Number analyzed (Participants) | 25
milliseconds/index | -1.94

4. Primary Outcome: Changes in Reaction Time as a Function of Theta Power.
Description: We measured the response time to auditory stimuli in milliseconds. We estimated EEG power using multitaper spectral analysis and calculated the power in decibels (dB) within the theta band (4 - 8 Hz).
Time Frame: Twenty minutes before the surgery.
Measure: Number; unit: milliseconds/decibels
Arm/Group | Study Group
Number analyzed (Participants) | 25
milliseconds/decibels | 30.11

ADVERSE EVENTS:
Time Frame: twenty minutes
Description: Adverse events are "any untoward or unfavorable medical occurrence including any abnormal sign, symptom or disease,...whether or not associated with the subject's participation in the research". Internal adverse events that are unexpected and related/possibly related to the research and external adverse events that are serious, unexpected and related/possibly related must be reported to the IRB within 5 working days/7 calendar days of the date the investigator first become aware of them.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=28)
Clinically significant respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Drop in blood oxygen saturation below 95%

LIMITATIONS AND CAVEATS:
We report these findings from a moderate-sized sample of subjects undergoing a structured protocol prior to general anesthesia. The sample size however is comparable and exceeds previous studies of fentanyl EEG effects. The EEG is commonly regarded as being noisy and prone to artifact, but in this clinical setting and with appropriate analyses methods we observed clear EEG signatures that correlated with predicted fentanyl effect site concentrations and with physiological and behavioral changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03866278/Prot_000.pdf